CLINICAL TRIAL: NCT01811745
Title: Physical Exercise and Jaques-Dalcroze Eurhythmics: Effects on Physical and Cognitive Functions, and Falls in Seniors (EPHYCOS Study)
Brief Title: Physical Exercise and Jaques-Dalcroze Eurhythmics: Effects on Physical and Cognitive Functions, and Falls in Seniors
Acronym: EPHYCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Andrea Trombetti, Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-175
Record Dates: First submitted 2013-03-12; First posted 2013-03-15 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Physical Function; Cognitive Function; Falls
Keywords: Aged; Cognition; Exercise; Falls; Gait; Physical function; Dual-task; Music; Postural Balance; Randomized controlled trial
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jaques-Dalcroze eurhythmics training (Experimental): Once-weekly 60-min Jaques-Dalcroze eurhythmics class, for 12 months.
  Interventions: Behavioral: Jaques-Dalcroze eurhythmics training
- Multicomponent exercise training (Active Comparator): Once-weekly 60-min multicomponent exercise class supplemented by one 30-min home-based exercise session, for 12 months.
  Interventions: Behavioral: Multicomponent exercise training

INTERVENTIONS:
Behavioral: Jaques-Dalcroze eurhythmics training — 12 months of weekly, supervised, structured, progressive, 60-min music-based multitask exercise classes (i.e., Jaques-Dalcroze eurhythmics). The music-based multitask program includes all exercises used in a previous work.
  Arms: Jaques-Dalcroze eurhythmics training
Behavioral: Multicomponent exercise training — 12 months of weekly, i) supervised, structured, progressive, 60-min multicomponent exercise classes, supplemented by ii) 30-min home-based exercise sessions. Briefly, the multimodal exercise program is based on core components for successful fall prevention in older adults. It contains balance, gait, coordination and strength training, with balance as a core component.
  Arms: Multicomponent exercise training

SUMMARY:
The purpose of this study is to evaluate the efficacy and the possible mechanisms underlying music-based multitask training (i.e., Jaques-Dalcroze eurhythmics) in older people, compared to multicomponent exercise training.

This study is designed as a 12-month, prospective, single-centre, single-blind, 2-arm, parallel group, randomized controlled trial in which 140 community-dwelling older adults at high risk of falls are randomly assigned to receive either a music-based multitask training intervention (i.e., Jaques-Dalcroze eurhythmics) or a multicomponent exercise training intervention, for 12 months. A 12-month follow-up is planned with outcome measures assessed at three time points: baseline (before intervention initiation), 6-month (intervention mid-point), and 12-month (intervention termination). Outcomes of interest include physical and cognitive performances, and falls. In addition, the investigators specifically address brain circuits in an exploratory sub-study. Volunteer trial participants from both study arms are invited to undergo functional magnetic resonance imaging (fMRI) at baseline and 12-month.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 65 years (no upper age limit)
* living in the community, even in protected housing
* identified as being at high risk of falls (i.e., one or more self-reported falls after the age of 65 years or balance impairment as assessed by a simplified Tinetti test or presence of one or two indicators of physical frailty based on Fried's criteria)
* willing to comply with all study requirements

Exclusion Criteria:

* neurological or orthopaedic disease (e.g., stroke with residual motor deficit, Parkinson's disease) with a significant impact on gait and balance performances
* fully dependent on a technical aid for walking such as canes or walker
* diagnosis of dementia based on a comprehensive neuropsychological assessment
* participation in a Jaques-Dalcroze Eurhythmics program or a supervised multicomponent exercise program in the past 12 months
* serious medical conditions or other factors that may limit adherence to interventions or affect conduct of the trial (e.g., terminal illness)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in gait variability under dual-task condition | 6 months, 12 months

SECONDARY OUTCOMES:
Change in gait performances (quantitative gait analysis under single and dual-task conditions) | 6 months, 12 months
Change in balance performances (quantitative balance analysis) | 6 months, 12 months
Change in functional tests performances (Timed Up & Go test and Short Physical Performance Battery) | 6 months, 12 months
Incidence of falls and fractures (prospective daily recording using calendars, to be returned monthly) | 6 months, 12 months
Change in cognitive performances (comprehensive neuropsychological battery assessing different aspects of executive functioning) | 6 months, 12 months
Change in anxiety/depression (Hospital Anxiety and Depression scale) | 6 months, 12 months
Change in fear of falling (Short-FESI) | 6 months, 12 months

OTHER OUTCOMES:
Change in brain networks (structural and functional levels) | 12 months
  fMRI sub-study

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Trombetti, MD, Principal Investigator — Bone Diseases Bone Diseases Service, Department of Internal Medicine Specialties, University Hospitals and Faculty of Medicine of Geneva
Locations (1):
- Bone Diseases Service, Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Background] Trombetti A, Hars M, Herrmann FR, Kressig RW, Ferrari S, Rizzoli R. Effect of music-based multitask training on gait, balance, and fall risk in elderly people: a randomized controlled trial. Arch Intern Med. 2011 Mar 28;171(6):525-33. doi: 10.1001/archinternmed.2010.446. Epub 2010 Nov 22. PMID 21098340